CLINICAL TRIAL: NCT00431899
Title: Effets of Fish Oil on Metabolic Fate of an Oral Glucose Load in Patients With End Stage Renal Disease Undergoing Hemodialysis
Brief Title: Effects of Omega 3 in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoire Régional de Nutrition Humaine (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HDW3
Record Dates: First submitted 2007-02-03; First posted 2007-02-06 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2007-02

CONDITIONS: Hemodialysis; End Stage Renal Disease
Keywords: nutrition; omega 3 fatty acids; insulin resistance
MeSH Terms: conditions — Kidney Failure, Chronic; Insulin Resistance

INTERVENTIONS:
Behavioral: fish oil supplementation

SUMMARY:
The aim of the study was to determine the effects of a 3-week fish oil oral supplementation on the metabolic fate and thermogenic effect of an oral glucose load in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis at least 6 months duration end stage renal disease

Exclusion Criteria:

* - Age < 18 y ou > 75 y
* Hemodialysis < 6 months
* Diabetes, obesity
* allergy to fish
* Asthma
* glucocorticoïds, propranolol,, Immunosuppressive drugs, Insulin, Somatostatin
* erythropoïetin < 3 months
* Cancer
* Hemoglobin < 11 g/l
* disease < 1 month
* pregnancy
* respiratory insufficiency
* intensive sport practice
* refusal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8
Dates: Start 2003-05; Study Completion 2003-11

PRIMARY OUTCOMES:
plasma glucose utilization
glucose-induced thermogenesis

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Delarue, MD,PhD, Principal Investigator — CHU Cavale Blanche F-29200 Brest
Locations (1):
- Laboratoire Régional de Nutrition Humaine, Brest, France